CLINICAL TRIAL: NCT00872690
Title: Factors Affecting Return to Work Among OEF/OIF Veterans With Polytrauma
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: D6661-R
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Trauma; Blast Injuries; Brain Injuries
Keywords: Multiple Trauma; Blast Injuries; Brain Injuries; Rehabilitation, Vocational; Consumer participation
MeSH Terms: conditions — Multiple Trauma; Blast Injuries; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: OEF/OIF veterans with polytrauma who have been referred by the Tampa VA Polytrauma Rehabilitation Center (PRC) to the VA VR&E Regional Office in St. Petersburg, Florida for Chapter 31 (IL) services.
- Group 2: Caregivers of the veterans who enroll in the study

SUMMARY:
The goal of this study is to examine things that make it easy or hard for OEF/OIF veterans with polytrauma to live independently or do things "on their own" at home and in the community.

DETAILED DESCRIPTION:
The Department of Veterans Affairs (VA) identifies employment as a priority issue for OEF/OIF veterans. However, OEF/OIF veterans with polytrauma represent a new and unique VA sub-population. Polytraumatic injuries are more complex than injuries sustained in any previous conflict. Returning to work, therefore, may prove especially challenging. Among individuals with severe disabilities, employment outcomes are closely tied to the individual's level of success with Independent Living (IL). IL refers to the ability to reside in the community and participate in activities of choice by managing available resources, negotiating barriers and exercising self-determination. IL often is viewed as a prerequisite to employment for severely disabled individuals, because barriers and facilitators to independence at home and in the community also influence success in the workplace. Thus, IL will be a critical first step to pursuing vocational/employment goals for OEF/OIF veterans with polytrauma. To date, no published studies have investigated IL among veterans with polytrauma. This pilot study will be the first project in a line of research to promote the independence and employability OEF/OIF veterans. The goals of the study are twofold. Goal 1 of the study is to investigate the barriers and facilitators to IL identified by community dwelling OEF/OIF veterans with polytrauma, caregivers, and IL service providers, and perceptions of how these factors may affect veterans' return to work. This goal will be accomplished by using qualitative methods for data collection and analyses. Qualitative interviewing will be used to elicit the perspectives of veterans with polytrauma and caregivers living in Florida, and Florida-based Vocational Rehabilitation and Employment IL service providers. Qualitative data will be coded, and then analyzed using the constant comparative method. Goal #2 of the study is to evaluate the feasibility of using the data collection tools and procedures for a future planned study. An efficacy evaluation will be used to test and refine the data collection tools (interview guides and demographic checklists). To evaluate data collection procedures, field notes will be recorded and analyzed to identify optimal organizational procedures and time parameters to minimize subject burden. Findings will be used to plan and design a large, national study of factors affecting return to work among OEF/OIF veterans with polytrauma living throughout the United States. Findings also will be used to develop future proposals to fund longitudinal research and implementation projects to improve employability outcomes among veterans with polytrauma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OEF/OIF related polytraumatic injuries

Exclusion Criteria:

* Polytraumatic injuries unrelated to OEF/OIF service

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Single, in-depth qualitative interviews | Single administration

SECONDARY OUTCOMES:
Demographic Checklist | Single administration

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M. Hannold, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (2):
- United States (2):
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida